CLINICAL TRIAL: NCT07324733
Title: Exploring the Novel Value of PSMA PET in Sjögren's Syndrome: Integrated Analysis With Established FAPI PET Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-PSS-PSMA
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Primary Sjögren Syndrome; PET

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pSS Dual-Tracer Imaging Arm (PSMA + FAPI PET) (Experimental): This arm includes patients diagnosed with primary Sjögren's syndrome. All participants undergo both PSMA PET and FAPI PET imaging. The PSMA PET scan is used to assess the functional integrity of salivary gland acinar cells, while the FAPI PET scan evaluates inflammatory and fibroblast activity within the same glands. The purpose of this arm is to characterize the functional-inflammatory relationship in pSS and to develop the combined PSMA/FAPI Index for disease staging and activity assessment.
  Interventions: Diagnostic Test: ⁶⁸Ga-PSMA PET/CT; Diagnostic Test: ⁶⁸Ga-FAPI PET/CT
- Prostate Cancer PSMA-Only Comparator Arm (Active Comparator): This arm consists of patients with prostate cancer who undergo PSMA PET imaging only, representing a population with preserved or physiologic salivary gland PSMA uptake. These scans serve as a reference group for establishing normal or baseline PSMA expression in salivary glands. This comparator arm allows differentiation between disease-related PSMA reduction in pSS and normal tracer distribution observed in patients without salivary gland pathology.
  Interventions: Diagnostic Test: ⁶⁸Ga-PSMA PET/CT

INTERVENTIONS:
Diagnostic Test: ⁶⁸Ga-PSMA PET/CT — PSMA PET imaging performed for clinical evaluation in prostate cancer patients, used as a comparator for physiologic salivary gland PSMA uptake.
Diagnostic Test: ⁶⁸Ga-FAPI PET/CT — FAPI PET imaging to assess inflammatory activity (FAPI) in patients with primary Sjögren's syndrome.
  Arms: pSS Dual-Tracer Imaging Arm (PSMA + FAPI PET)

SUMMARY:
Primary Sjögren's syndrome (pSS) is a chronic autoimmune exocrinopathy characterized by lymphocytic infiltration, progressive destruction of salivary gland acini, and varying degrees of functional impairment and fibrosis. Conventional imaging provides limited ability to simultaneously evaluate glandular function and inflammatory activity, leading to challenges in disease staging and treatment decision-making. This study explores a conceptual dual-tracer imaging framework using PSMA PET and FAPI PET to delineate complementary biological processes in pSS.

DETAILED DESCRIPTION:
Based on current evidence, salivary gland acinar cells physiologically express PSMA; thus, reduced PSMA uptake may reflect loss of functional parenchyma in patients with pSS. In contrast, activated fibroblasts markedly express FAP, and increased FAPI uptake correlates with ongoing inflammation and fibroblast-driven remodeling. We hypothesize that within the same gland, functional decline (PSMA↓) and inflammatory activity (FAPI↑) may coexist and exhibit a negative correlation, forming a paired imaging biomarker that captures both pathological dimensions. By integrating these two signals into a combined PSMA/FAPI Index, this approach may enable more precise characterization of the "function-inflammation" spectrum in pSS, providing a noninvasive tool for disease staging, monitoring, and potentially predicting therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Fulfillment of the 2016 ACR-EULAR Classification Criteria for pSS at enrollment. OR diagnosis of a solid tumor scheduled for FAPI PET imaging

Exclusion Criteria:

* Combined with tumors or other connective tissue diseases (for SS group);
* Patients who are currently using hormones/biological agents (for both groups)；
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Salivary Gland PSMA Uptake Across Groups | Baseline
  Quantitative comparison of PSMA PET uptake parameters (SUVmax, SUVmean) of the parotid glands among three groups: pSS patients, individuals with normal salivary glands, and prostate cancer patients.

SECONDARY OUTCOMES:
Multiglandular PSMA Uptake Comparison | Baseline
  Evaluation of PSMA PET uptake (SUVmax, SUVmean) in the parotid, submandibular, and lacrimal glands across the same study groups.
Correlation Between PSMA Uptake and Clinical Indicators | Baseline
  Correlation of salivary gland PSMA SUV values with clinical, immunological, and functional markers of pSS, including ESR, CRP, IgG, RF, anti-SSA/SSB titers, unstimulated whole salivary flow rate, sialography findings, ESSDAI, and ESSPRI scores.
Quantitative and Spatial Relationship Between PSMA and FAPI Uptake Definition | Baseline
  1. Quantitative correlation: Association between PSMA SUV and FAPI SUV in the same glands.
  2. Spatial co-localization: Overlap or complementarity of low-PSMA and high-FAPI regions within individual glands using image fusion and voxel-based analysis (e.g., Dice coefficient).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China